CLINICAL TRIAL: NCT03903523
Title: Efficacy and Safety of Lumen Apposing Metal Stents: a Retrospective Multicentre Study
Brief Title: Efficacy and Safety of Lumen Apposing Metal Stents
Acronym: LAMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 970
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Biliary Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Lumen apposing metal stent (LAMS) — Stent positioning

SUMMARY:
Endoscopic ultrasonography (EUS) has revolutioned the management of gastroenterological patients and is acquiring an increasingly important role.

The development of specifically designed stents has significantly increased the technical and clinical success rate of the EUS-guided procedures, considerably reducing the rate of adverse events. Currently EUS has a prominent role in drainage of peripancreatic fluid collections and it represents an important therapeutic option for patients with distal malignant biliary obstruction, in which the ERCP fails, allowing the positioning of a transgastric or transbulbar lumen apposing metal stent (LAMS) to drain the biliary duct. Moreover, the EUS-guided gallbladder drainage of patients with high surgical risk and acute cholecystitis, which cannot be operated, is another important therapeutic indication.

Our aim is to perform a multicentre retrospective analysis of all types of EUS drainage (gallbladder drainage, biliary drainage, peripancreatic fluid collection drainage) with the positioning of LAMS in order to evaluate the rate of technical and clinical success and to assess the safety profile of these procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients with distal malignant common bile duct obstruction with failed ERCP
* Patients with symptomatic peripancreatic fluid collections
* Patients with acute cholecystitis who are unfit for surgery
* Agree to receive follow up phone calls
* Able to provide written informed consent

Exclusion Criteria:

* Coagulation and/or platelets hereditary disorders.
* Pregnant women
* Inability to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective analysis of a prospectively maintained database of all consecutive patients with distal malignat biliary obstruction, high surgical risk acute cholecystitis, or symptomatic pancreatic fluid collection that underwent EUS drainage from January 2016 to December 2022. All EUS drainage were performed by experienced operators.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-04-30 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the rate of technical and clinical success of EUS drainage (gallbladder drainage, biliary drainage, peripancreatic fluid collection drainage) with the positioning of lumen apposing metal stents | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Anderloni, MD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (2):
- Italy (2):
  - Endoscopy Unit, Humanitas Research Hospital, Rozzano, Milano
  - Humanitas Research Hospital, Milan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Binda C, Anderloni A, Fugazza A, Amato A, de Nucci G, Redaelli A, Di Mitri R, Cugia L, Pollino V, Macchiarelli R, Mangiavillano B, Forti E, Brancaccio ML, Badas R, Maida M, Sinagra E, Repici A, Fabbri C, Tarantino I. EUS-guided gallbladder drainage using a lumen-apposing metal stent as rescue treatment for malignant distal biliary obstruction: a large multicenter experience. Gastrointest Endosc. 2023 Nov;98(5):765-773. doi: 10.1016/j.gie.2023.06.054. Epub 2023 Jun 29. PMID 37392954
- [Derived] Fugazza A, Fabbri C, Di Mitri R, Petrone MC, Colombo M, Cugia L, Amato A, Forti E, Binda C, Maida M, Sinagra E, Repici A, Tarantino I, Anderloni A; i-EUS Group. EUS-guided choledochoduodenostomy for malignant distal biliary obstruction after failed ERCP: a retrospective nationwide analysis. Gastrointest Endosc. 2022 May;95(5):896-904.e1. doi: 10.1016/j.gie.2021.12.032. Epub 2022 Jan 4. PMID 34995640
- [Derived] Facciorusso A, Amato A, Crino SF, Sinagra E, Maida M, Fugazza A, Binda C, Coluccio C, Repici A, Anderloni A, Tarantino I, Fabbri C; i-EUS Group. Definition of a hospital volume threshold to optimize outcomes after drainage of pancreatic fluid collections with lumen-apposing metal stents: a nationwide cohort study. Gastrointest Endosc. 2022 Jun;95(6):1158-1172. doi: 10.1016/j.gie.2021.12.006. Epub 2021 Dec 18. PMID 34932991